CLINICAL TRIAL: NCT07069348
Title: The Bearing Between Systemic Lupus Erythematosus Severity With Vitamin D Through Treg Cell Entanglement in Pediatric Patients
Brief Title: SLE Severity Linked to Vitamin D Via Treg Cells in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Wisnu Barlianto (Other)
Responsible Party: Sponsor-Investigator, Wisnu Barlianto, Prof. Dr. dr. WISNU BARLIANTO, M.Si.Med., Sp.A(K)., University of Brawijaya
Organization: University of Brawijaya (Other)
Other Study IDs: SLE VIT D Treg
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: SLE

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SLE ped: SLE pediatric patients without intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — There is no treatment or intervention administered to the patients

SUMMARY:
SLE has been characterized by dysfunctional or decreased numbers of Treg cells because one of it function is to prevent autoimmunity. Vitamin D has already known to increase the number and function of Treg by enhancing their differentiation and expansion. This study aims to investigate the relationship between SLE severity in pediatric patients and vitamin D levels through modulation of Treg cells. This is a cross-sectional study of all children aged 7-18 years old who sought care for SLE at Dr. Saiful Anwar Hospital Malang between March 2024 until December 2024. 25(OH)D level was obtained by ELISA, Treg cell percentage was obtained by flow cytometry, and patient severity was measured by SLEDAI score.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a chronic autoimmune disease that affects multiple organ systems and often begins during childhood or adolescence. Regulatory T cells (Treg) play a critical role in suppressing autoimmune responses, and several studies have shown that patients with SLE tend to have reduced numbers and/or function of Treg cells. Vitamin D has been reported to enhance Treg cell differentiation and function, suggesting a potential immunomodulatory role.

This cross-sectional observational study aims to evaluate the relationship between vitamin D status and disease severity in pediatric patients with SLE by examining the role of Treg cells as a potential mediator. Pediatric patients aged 7 to 18 years who are diagnosed with SLE and receiving care at Dr. Saiful Anwar Hospital, Malang, between March and December 2024 will be included. Serum 25(OH)D levels will be measured using ELISA, and Treg cell percentages will be assessed via flow cytometry. Disease severity will be determined using the SLE Disease Activity Index (SLEDAI).

Findings from this study are expected to provide insight into the immunological mechanism involving vitamin D and Treg cells in pediatric SLE and potentially guide future interventions or supplementation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 7 to 18 years.
* Diagnosed with Systemic Lupus Erythematosus (SLE) based on ACR or SLICC classification criteria.
* Receiving care or follow-up at Dr. Saiful Anwar Hospital, Malang during the study period and willing to participate in the study and provide informed consent (from parents or guardians).

Exclusion Criteria:

* Currently receiving vitamin D supplementation or medications known to influence vitamin D metabolism (e.g., anticonvulsants, glucocorticoids in high doses, etc.).
* Diagnosed with chronic kidney disease, liver disease, or malabsorption disorders.
* Diagnosed with other autoimmune diseases besides SLE.
* Presence of acute infection or fever at the time of data collection.
* Incomplete clinical or laboratory data required for analysis (e.g., missing ELISA or flow cytometry results).

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients aged 7 to 18 years who have been diagnosed with Systemic Lupus Erythematosus (SLE) and are receiving care at Dr. Saiful Anwar Hospital, Malang, Indonesia. Participants are recruited between March and December 2024 as part of a cross-sectional observational study evaluating vitamin D levels, Treg and Th17 cell percentage, zinc serum, and disease severity.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

PRIMARY OUTCOMES:
25-hydroxyvitamin D (25(OH)D) | At the time of enrollment
  Correlation between serum 25(OH)D levels and SLE disease activity (SLEDAI score)
Zinc serum | At the time of enrollment
  Correlation between Zinc serum and SLE disease activity (SLEDAI score)
The Percentage of Th17 and Treg | At the time of enrollment
  Correlation between The Percentage of Th17 and Treg with SLE disease activity (SLEDAI score)

CONTACTS AND LOCATIONS:
Overall Officials: Wisnu Barlianto, Prof., Study Chair — Faculty of Medicine Universitas Brawijaya
Locations (1):
- Universitas Brawijaya, Malang, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
We will maintain the confidentiality of our patients' data